CLINICAL TRIAL: NCT03918005
Title: Effects of Hypocaloric Diets With Different Glycemic Loads on Pulse Wave Velocity in Overweight and Obese Adults: a Randomized Clinical Trial
Brief Title: Effects of Hypocaloric Diets With Different Glycemic Loads on Pulse Wave Velocity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Lisiane Perin, Principal Investigator, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lisianeperin@hotmail.com
Record Dates: First submitted 2019-04-02; First posted 2019-04-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Glycemic Index; Overweight; Obesity; Pulse Wave Velocity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low glycemic load diet (Experimental): Foods with low glycemic index or glycemic load (brown rice, brown bread, whole wheat pasta, oat bran, yogurt, milk, apple, pear, peach)
  Interventions: Other: Low glycemic load diet
- High glycemic load diet (Active Comparator): Foods with high glycemic index or glycemic load (white rice, white bread, corn flakes, mashed potatoes, orange juice, banana, persimmon, grape, raisins, honey, sugar)
  Interventions: Other: Low glycemic load diet

INTERVENTIONS:
Other: Low glycemic load diet — Foods with low glycemic index or glycemic load (brown rice, brown bread, whole wheat pasta, oat bran, yogurt, milk, apple, pear, peach)

SUMMARY:
Worldwide, in terms of attributable deaths, the main intermediate risk factor for the development of cardiovascular diseases is systemic arterial hypertension, followed by overweight and sustained hyperglycemia. These factors have positively influenced public and private spending on health. The more robust studies showed that age is one of the main determinants of arterial stiffness. However, there is a possibility that other variables, such as elevated glucose levels, obesity, and systemic inflammation itself, as well as insulin resistance are important factors in this scenario. On the other hand, the measurement of the pulse wave velocity is widely acceptable for the evaluation of the arterial stiffness, inferring the cardiovascular risk in different populations. Since arterial stiffness is influenced by hemodynamic forces and inflammatory mediators, which may be related to sodium and glucose balance, it is necessary to evaluate whether a hypocaloric and low glycemic load diet, in a thesis that decreases lipid and inflammatory levels, may have favorable effects on pulse wave velocity in overweight adults.

DETAILED DESCRIPTION:
The diets will be calculated in Microsoft Excel 2018 software, using tables of nutritional composition, glycemic index and glycemic load, which have foods with high glycemic index or glycemic load (white rice, white bread, corn flakes, mashed potatoes, orange juice (brown rice, whole wheat bread, whole noodles, oat bran, yogurt, milk, apple, pear, peach). The methodology for calculating GC estimates will be based on the FAO / WHO Protocol. The diets will be designed in 1200, 1400, 1600, 1800 and 2000 kcal / day. All participants will be categorized according to one of the five levels of the diet's energy content. In addition, all patients will receive a leaflet with nutritional guidelines according to their diet.

During the study, participants will be required to maintain their medication consumption, if any, as prescribed by a physician. To assess adherence to the diet, participants will consult with a nutritionist on a weekly basis and complete the 24-hour food recall.

It will be measured the pulse wave velocity.This outcome will be evaluated before the beginning of the diets and 6 weeks after the beginning of the diets.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Between 20 and 59 years old
* Body mass index ≥ 25.0 kg/m²
* Physically inactive (physical activity <150 min/week)

Exclusion Criteria:

* Pregnant women
* Vegetarians
* Vegans
* Users of dietary supplements
* Smokers
* Alcohol abusers (men: more than 4 doses in a single day or more than 14 doses per week; women: more than 3 doses in a single day or more than 7 doses per week)
* Individuals with a previous diagnosis of hypertension
* Chronic kidney disease
* Type 1 or 2 diabetes mellitus
* Hypothyroidism
* Hyperthyroidism
* Events in the last 6 months (coronary artery disease, acute myocardial infarction, cerebral vascular disease, peripheral arterial disease, or heart failure)

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 92 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | 6 weeks
  The calibrated and validated Mobil-O-Graph® portable monitor (IEM GmbH, Stolberg, Germany) will be used. This module is connected to a computer to record the brachial pulse wave. It performs pulse wave analysis based on the oscillometric method. The arterial pulsation generates pressure oscillations, which are transmitted to the blood pressure cuff and measured by the transducer to be interpreted by a specific software, recording the pulse wave of the brachial artery and deriving a pulse wave from the aortic arch.
  All measurements will be performed by the same evaluator on the right side of the volunteer, at rest. Subjects will be instructed to be with empty bladder, not to drink coffee 60 minutes before gauging and alcoholic beverage in the last 24 hours.
  The pulse wave velocity will be evaluated before the beginning of the diets and 6 weeks after the beginning of the diets.

CONTACTS AND LOCATIONS:
Overall Officials: Lisiane Perin, MsC, Principal Investigator — Instituto de Cardiologia / Fundação Universitária de Cardiologia

IPD SHARING:
Plan to Share IPD: No